CLINICAL TRIAL: NCT03436732
Title: A Phase I Study of the Mesothelin-Targeted Immunotoxin LMB-100 in Combination With SEL-110 in Subjects With Malignant Pleural or Peritoneal Mesothelioma
Brief Title: Mesothelin-Targeted Immunotoxin LMB-100 in Combination With SEL-110 in Subjects With Malignant Pleural or Peritoneal Mesothelioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to fatal occurrence (pneumonitis) attributed to one of the study drugs.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180057; 18-C-0057
Record Dates: First submitted 2018-02-16; First posted 2018-02-19 (Actual); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Mesothelioma
Keywords: Immunotoxin; Rapamycin; Targeted Therapy; Mesothelin
MeSH Terms: conditions — Mesothelioma | interventions — LMB-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Dose Escalation (Experimental): Dose escalation - patients with mesothelioma treated with LMB-100+SEL-110 at escalating doses
  Interventions: Drug: LMB-100; Drug: SEL-110
- 2/Dose Expansion (Experimental): Dose expansion - patients with mesothelioma treated with LMB-100+SEL-110 at recommended phase 2 dose (RP2D)
  Interventions: Drug: LMB-100; Drug: SEL-110

INTERVENTIONS:
Drug: LMB-100 — administered on days 1, 3 and 5 of each 21 day cycle for up to 4 cycles
Drug: SEL-110 — administered on day 1 of each cycle for up to 4 cycles

SUMMARY:
Background:

Mesothelioma is cancer of the tissue that lines some organs. A new drug, LMB-100, may bind to a protein on mesothelioma tumors and kill cancer cells. But sometimes the body makes antibodies that reduce how well LMB-100 works. Researchers want to see if adding the drug SEL-110 to LMB-100 will prevent these antibodies from forming.

Objective:

To learn how safe and tolerable LMB-100 plus SEL-110 is in people with advanced mesothelioma.

Eligibility:

Adults ages 18 and older who have pleural or peritoneal mesothelioma that has not responded to prior platinum-based therapy

Design:

Participants will be screened with

* Medical history
* Physical exam
* Blood and urine tests
* Sample of tumor tissue. This can be from a previous procedure.
* Scan of the chest, abdomen, and pelvis. Participants will lie on a table in a scanner that takes pictures. A special dye may be injected in a vein.
* Positron emission tomography (fludeoxyglucose positron emission tomography (FDG-PET)) scan. A sugar attached to a chemical that gives off a signal will be injected before the scan.
* Heart function tests

The study will be done in 21-day cycles. Participants will get the study drugs for up to 4 cycles. They will get them through an intravenous (IV) catheter (a tube inserted in a vein, usually in the arm):

* LMB-100 for about 30 minutes on day 1, day 3, and day 5 of each cycle
* SEL-110 for about 1 hour on day 1 of each cycle

Participants will get standard medicines to help prevent side effects.

Participants will repeat some screening tests during each cycle and about 5 weeks after the last dose of study drug.

DETAILED DESCRIPTION:
Background:

* LMB-100 and a closely related immunotoxin also targeting mesothelin have been studied in previous Phase 1 clinical studies for mesothelioma and pancreatic cancer.
* Results from these studies showed that the majority of patients formed anti-drug-antibodies (ADAs) that neutralized subsequent injection of the product making it ineffective.
* In a small subset of patients that did not form ADAs to the product, good response and regression of tumors was seen.
* In a different application SEL-110, a biodegradable nanoparticle containing rapamycin, has been shown in clinical trials to prevent the formation of ADAs to an immunogenic enzyme when co-administered. Preclinical data show that SEL-110 also prevents the formation of ADAs to LMB-100.
* This clinical trial will investigate whether SEL-110 when administered with LMB-100 is able to prevent the formation of ADAs and thus allow patients to receive multiple, effective injections of LMB-100.

Objectives:

-The primary objective of the study is to assess the safety and tolerability of LMB-100 in combination with SEL-110.

Eligibility:

Primary Inclusion Criteria

* Greater than or equal to 18 years of age
* Histologically confirmed epithelial or biphasic pleural or peritoneal mesothelioma not amenable to potentially curative surgical resection.
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients must have had at least one prior chemotherapy regimen that includes pemetrexed and cisplatin or carboplatin. There is no limit to the number of prior chemotherapy regimens received.
* Patients for whom no standard curative therapy exists

Primary Exclusion Criteria:

* Known or clinically suspected central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases.
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results.
* Evidence of active or uncontrolled infections.
* Live attenuated vaccinations 14 days prior to treatment
* Pregnant women are excluded from this study

Design:

* This is a Phase I, single center, dose escalation study of LMB-100 in combination with SEL-110
* Patients will receive the combination using a dose escalation scheme in which different doses of LMB100 and SEL-110 will be evaluated.
* Patients will receive 4 cycles of LMB-100 with SEL-110. A cycle will consist of intravenous (i.v.) infusion of SEL-110 on Day 1 of the cycle followed immediately by an i.v. infusion of LMB-100, then on Days 3 and 5 of the cycle patients will receive an i.v. infusion of LMB-100 only. Treatment cycles will be separated by 21 days.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically confirmed epithelial or biphasic pleural or peritoneal mesothelioma not amenable to potentially curative surgical resection. However, patients with biphasic tumors that have a more than or equal to 50% sarcomatoid component will be excluded.

The diagnosis will be confirmed by the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI).

* Archival sample or fresh biopsy or tumor effusion must be available for confirmation of diagnosis.
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients must have had at least one prior chemotherapy regimen that includes pemetrexed and cisplatin or carboplatin. There is no limit to the number of prior chemotherapy regimens received.
* The last dose of previous therapy must have occurred at least 3 weeks prior to the start of study therapy. Palliative radiotherapy is allowed up to 2 weeks before the first LMB-100 infusion.
* Patients for whom no standard curative therapy exists
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of LMB-100 + SEL-110 in patients <18 years of age, children are excluded from this study
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade less than or equal to 1, except alopecia (any grade) and Grade 2 peripheral neuropathy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Adequate hematological function: neutrophil count of more than or equal to 1.0 times 10(9) cells/L, platelet count of greater than or equal to 100,000/mcL, hemoglobin more than or equal to 9 g/dL
* Adequate liver function: Bilirubin less than or equal to 2.5 times the upper limit of normal (ULN) (excluding Gilbert's Syndrome, see below).
* Patients with Gilbert's syndrome will be eligible for the study. The diagnosis of Gilbert's syndrome is suspected in people who have persistent, slightly elevated levels of unconjugated bilirubin without any other apparent cause. A diagnosis of Gilbert's syndrome will be based on the exclusion of other diseases based on the following criteria:

  1. Unconjugated hyperbilirubinemia noted on several occasions
  2. No evidence of hemolysis (normal hemoglobin, reticulocyte count, and lactate dehydrogenase (LDH))
  3. Normal liver function tests
  4. Absence of other diseases associated with unconjugated hyperbilirubinemia
* Adequate renal function: creatinine clearance (by Cockcroft Gault formula) greater than or equal to 50 mL/min.
* Must have serum albumin > 2.5 g/dL without intravenous supplementation
* Must have left ventricular ejection fraction > 50%
* Must have an ambulatory oxygen saturation of > 90% on room air
* The effects of LMB-100 in combination with SEL-110 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry until 3 months after the last dose of study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Known or clinically suspected central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases. History or clinical evidence of CNS metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days.
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including significant pulmonary disease other than primary cancer, uncontrolled diabetes mellitus, and/or significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, uncontrolled arrhythmias, unstable angina, non-compensative congestive heart failure, or clinically significant pericardial effusion)
* Active or uncontrolled infections.
* Human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. HIV positive patients will be excluded due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.
* Patients with prior pneumonectomy
* Prior therapy with LMB-100
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury greater than or equal to 28 days prior to the first LMB-100 infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Dementia or altered mental status that would prohibit informed consent
* Live attenuated vaccinations 14 days prior to treatment
* Pregnant women are excluded from this study because it is unknown whether LMB-100 + SEL 100 has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100+SEL-110, breastfeeding should be discontinued if the mother is treated with LMB-100+SEL-110. These potential risks may also apply to other agents used in this study.
* Known hypersensitivity to any of the components of LMB-100 and/or SEL-110
* Presence of immunosuppressive conditions, including administration of any medications or treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids (oral or injectable) during 3 months prior to enrollment.

Inhaled and topical corticosteroids allowed.

* Known allergy to polyethylene glycol (PEG)ylated products.
* History of anaphylactic reaction to a recombinant protein or hypersensitivity to PEG.
* Taken an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study.
* Taken a strong inhibitor or inducer of cytochrome P450 3A4 (CYP3A4) within 14 days prior to enrollment (see Flockhart Table or similarly updated source for a list of such agents)
* Taken drugs known to interact with Rapamune such as cyclosporine, diltiazem, erythromycin, ketoconazole (and other antifungals), nicardipine (and other calcium channel blockers), rifampin, verapamil within 14 days prior to enrollment
* Uncontrolled hypertension (above 150/95 mm Hg).
* History of end-stage renal disease requiring dialysis.
* Serum phosphorus less than 2.0 mg/dL
* Organ transplant recipient

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0057.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1/5 participants enrolled was a screen failure following enrollment.
Groups:
- 140 mcg/kg LMB-100 + SEL-110; 100 mcg/kg LMB-100 + SEL-110: Dose escalation - patients with mesothelioma treated with LMB-100+SEL-110 at escalating doses
  LMB-100: administered on days 1, 3 and 5 of each 21 day cycle for up to 4 cycles
  SEL-110: administered on day 1 of each cycle for up to 4 cycles
Period: Overall Study
Arm/Group | 140 mcg/kg LMB-100 + SEL-110 | 100 mcg/kg LMB-100 + SEL-110
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Not treated-enrolled in different study | 1 | 0
Not completed — Off study after cycle 1 | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 140 mcg/kg LMB-100 + SEL-110 | 100 mcg/kg LMB-100 + SEL-110 | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.75 (2.278) | 58 (0) | 63 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade ≥3 Adverse Events Related to Study Drug at Dose Level 140 mcg/kg and 100 mcg/kg
Description: Here are the grade ≥3 adverse events at each dose level assessed by the Common Terminology Criteria in Adverse Events CTCAE v5.0. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is Severe or medically significant but not immediately life-threatening;hospitalization or prolongation of hospitalization indicated; disabling;limiting self care ADL (i.e., bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden. Grade 4 is life-threatening consequences;urgent intervention indicated. Grade 5 is death related to adverse event.
Time Frame: Day 85
Measure: Count of Participants; unit: Participants
Groups:
- 140 mcg/kg; 100 mcg/kg: Dose escalation - patients with mesothelioma treated with LMB-100+SEL-110 at escalating doses
  LMB-100: administered on days 1, 3 and 5 of each 21 day cycle for up to 4 cycles
  SEL-110: administered on day 1 of each cycle for up to 4 cycles
Arm/Group | 140 mcg/kg | 100 mcg/kg
Number analyzed (Participants) | 4 | 1
Participants
  Grade 4 pericardial effusion | 1 | 0
  Grade 5 pneumonitis | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the highest tested dose of LMB-100 and SEL-110 at which no more than 1 of 6 subjects experience a dose limiting toxicity. A dose limiting toxicity is defined as any of the following: Grade 4 neutropenia for a minimum duration of 7 days. Grade 4 thrombocytopenia (≤25.0 x 10(9) cells/L), Grade 3 thrombocytopenia associated with bleeding episodes, and Grade 4 anemia. Grade ≥3 non-hematological toxicity with the exception of Alopecia (any grade), Grade 3 nausea and vomiting lasting > 48 hours despite appropriate treatment, Grade 3 diarrhea lasting for ≤ 2 days with no fever or dehydration, and laboratory values of ≥ grade 3 that are judged not clinically significant by the investigator. Any other drug related toxicity considered significant enough to be qualified as a DLT in the opinion of the principal investigator. Inability to start cycle 2 within 3 weeks after completing cycle 1 due to drug-related adverse events.
Time Frame: Day 21
Population: MTD was not found because the study was closed due to a fatal occurrence of pneumonitis that was attributed to one of the study drugs.
Arm/Group | 1/Dose Escalation
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Partial Response or Complete Response (PR + CR)
Description: Response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesion, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | 140 mcg/kg | 100 mcg/kg
Number analyzed (Participants) | 4 | 1
Participants
  Partial Response | 0 | 0
  Complete Response | 0 | 0

4. Secondary Outcome: Fraction of Participants With Detectable LMB-100 in Blood After Cycle 4
Description: Blood is measured for a detectable level of LMB-100 in the blood. LMB-100 is either detectable in the blood or not. A detectable level of LMB-100 in the blood is considered a desirable outcome for the participant. Hence, the reverse is not a considered a desirable outcome for the participant.
Time Frame: Day 85
Population: This outcome measure was not done because the study was closed due to a fatal occurrence of pneumonitis that was attributed to one of the study drugs.
Arm/Group | 140 mcg/kg | 100 mcg/kg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately one month and 25 days for the 100 mcg/kg Arm/Group, and 9 months and 28 days for the 140 mcg/kg Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | 140 mcg/kg | 100 mcg/kg
Number analyzed (Participants) | 4 | 1
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately one month and 25 days for the 100 mcg/kg Arm/Group, and 9 months and 28 days for the 140 mcg/kg Arm/Group.
Arm/Group | 140 mcg/kg LMB-100 + SEL-110 | 100 mcg/kg LMB-100 + SEL-110
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/1
Other Adverse Events (participants affected / at risk) | 3/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 140 mcg/kg LMB-100 + SEL-110 (N=4) | 100 mcg/kg LMB-100 + SEL-110 (N=1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Death
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (3) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 140 mcg/kg LMB-100 + SEL-110 (N=4) | 100 mcg/kg LMB-100 + SEL-110 (N=1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
CPK increased (Investigations) | 1 (2) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Edema face (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 1 (3)
Fatigue (General disorders) | 1 (1) | 1 (2)
Fever (General disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, Chest discomfort (General disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 1 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (6) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (9) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (12) | 1 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Weight gain (Investigations) | 2 (2) | 1 (5)
Weight loss (Investigations) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03436732/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03436732/ICF_001.pdf